CLINICAL TRIAL: NCT02367118
Title: Prednisone in Chronic Rhinosinusitis Without Nasal Polyps. A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Prednisone in Chronic Rhinosinusitis Without Nasal Polyps
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Sociedad Chilena de Otorrinolaringología, Medicina y Cirugía de Cabeza y Cuello (Unknown)
Responsible Party: Principal Investigator, Constanza J. Valdes, MD, Professor Assistant University of Chile. Department of Otorhinolaryngology-Head and Neck Surgery., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRD- CRSsNP-1
Record Dates: First submitted 2015-02-08; First posted 2015-02-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Sinusitis; Chronic Rhinosinusitis
Keywords: chronic rhinosinusitis without nasal polyps prednisone
MeSH Terms: conditions — Sinusitis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Experimental): Intervention: prednisone 5 mg tablets taken orally, in decreasing doses. Beginning with 6 tablets (30 mg) daily for 7 days, then 3 tablets (15 mg) daily for 7 days, then 1 tablet (5 mg) daily for 7 days. Total days of treatment: 21 days.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Intervention: placebo tablets taken orally (similar to prednisone), in decreasing doses. Beginning with 6 tablets daily for 7 days, then 3 tablets daily for 7 days, then 1 tablet daily for 7 days. Total days of treatment: 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone
  Arms: Prednisone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether prednisone is effective in the treatment of chronic rhinosinusitis without nasal polyps in adult patients.

DETAILED DESCRIPTION:
General Objective:

1. Compare clinical improvement in adult patients with chronic rhinosinusitis without nasal polyps (CRSsNP) through application of SNOT 22 questionnaire and visual analogue scale of symptoms, sniff test, acoustic rhinometry and rhinomanometry and nasal endoscopy using Lund-Kennedy score, after 6 months of follow-up after treatment prednisone or placebo plus standard medical treatment for 21 days.

Specific Objectives:

1. Compare decreased in SNOT-22 questionnaire score and visual analog scale of symptoms after treatment with prednisone or placebo.
2. Compare decreased in nasal endoscopy findings, through application of Lund-Kennedy score, after treatment with prednisone or placebo.
3. Compare improvements in smell after treatment with prednisone or placebo.
4. Determine whether there are differences in nasal permeability measured by rhinomanometry and acoustic rhinometry after treatment with prednisone or placebo.
5. Determine whether there is a difference in the SNOT 22 questionnaire score, visual analogue scale of symptoms, score of smell and Lund-Kennedy score between CRSsNP patients and eosinophilia, and CRSsNP patients with normal eosinophils, receiving prednisone or placebo .
6. Determine if there is a difference in the SNOT 22 questionnaire score, visual analogue scale of symptoms, score of smell and Lund-Kennedy score between CRSsNP patients with elevated total immunoglobulin E and CRSsNP patients with normal total immunoglobulin E, receiving treatment with prednisone or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRSsNP as recommended European Position Paper on Rhinosinusitis and Nasal Polyps 2012

Exclusion Criteria:

* Treatment with oral corticosteroids or topical corticosteroids the last 4 weeks.
* Previous surgical treatment for CRSsNP
* History of diabetes mellitus and / or glaucoma and / or decompensated hypertension and / or gastric ulcer.
* Pregnancy.
* History of cystic fibrosis, primary ciliary dyskinesia, immunodeficiency, allergic fungal sinusitis, nasal polyps, nasal tumors, hepatic or renal dysfunction.
* Hypersensitivity to prednisone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Symptoms as measured by SNOT 22 questionnaire and visual analogue scale at 6 months | Improvement in symptoms at the end (average of 25 days is expected) of the administration of prednisone (intervention), one month, three months and six months after the end of intervention compared to placebo
Change in Olfactory function as measured by "Sniffin'Sticks 12 tests" at 6 months | Improvement in Olfactory function at the end (average of 25 days is expected) of the administration of prednisone (intervention), one month, three months and six months after the end of intervention compared to placebo
Change in Nasal patency as measured by Acoustic rhinometry and Rhinomanometry at 6 months | Improvement in nasal patency at the end (average of 25 days is expected) of the administration of prednisone (intervention), one month, three months and six months after the end of intervention compared to placebo
Changes in Nasal endoscopy findings as measured by Lund-Kennedy score at 6 months | Changes in nasal endoscopy findings at the end (average of 25 days is expected) of the administration of prednisone (intervention), one month, three months and six months after the end of intervention compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Constanza J Valdes, MD, Study Director — University of Chile; Marcela A Veloz, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital del Salvador, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Bhattacharyya N, Orlandi RR, Grebner J, Martinson M. Cost burden of chronic rhinosinusitis: a claims-based study. Otolaryngol Head Neck Surg. 2011 Mar;144(3):440-5. doi: 10.1177/0194599810391852. Epub 2011 Feb 3. PMID 21493210
- [Background] Dubin MG, Liu C, Lin SY, Senior BA. American Rhinologic Society member survey on "maximal medical therapy" for chronic rhinosinusitis. Am J Rhinol. 2007 Jul-Aug;21(4):483-8. doi: 10.2500/ajr.2007.21.3047. PMID 17882920
- [Background] Mullol J, Obando A, Pujols L, Alobid I. Corticosteroid treatment in chronic rhinosinusitis: the possibilities and the limits. Immunol Allergy Clin North Am. 2009 Nov;29(4):657-68. doi: 10.1016/j.iac.2009.07.001. PMID 19879441
- [Background] Takeda K, Takeno S, Hirakawa K, Ishino T. Expression and distribution of glucocorticoid receptor isoforms in eosinophilic chronic rhinosinusitis. Auris Nasus Larynx. 2010 Dec;37(6):700-7. doi: 10.1016/j.anl.2010.03.005. Epub 2010 May 21. PMID 20488636
- [Background] Benitez P, Alobid I, de Haro J, Berenguer J, Bernal-Sprekelsen M, Pujols L, Picado C, Mullol J. A short course of oral prednisone followed by intranasal budesonide is an effective treatment of severe nasal polyps. Laryngoscope. 2006 May;116(5):770-5. doi: 10.1097/01.mlg.0000205218.37514.0f. PMID 16652085
- [Background] Lund VJ, Kennedy DW. Quantification for staging sinusitis. The Staging and Therapy Group. Ann Otol Rhinol Laryngol Suppl. 1995 Oct;167:17-21. PMID 7574265
- [Background] Kobal G, Klimek L, Wolfensberger M, Gudziol H, Temmel A, Owen CM, Seeber H, Pauli E, Hummel T. Multicenter investigation of 1,036 subjects using a standardized method for the assessment of olfactory function combining tests of odor identification, odor discrimination, and olfactory thresholds. Eur Arch Otorhinolaryngol. 2000;257(4):205-11. doi: 10.1007/s004050050223. PMID 10867835
- [Background] Poetker DM, Reh DD. A comprehensive review of the adverse effects of systemic corticosteroids. Otolaryngol Clin North Am. 2010 Aug;43(4):753-68. doi: 10.1016/j.otc.2010.04.003. PMID 20599080
- [Background] Heinzerling L, Mari A, Bergmann KC, Bresciani M, Burbach G, Darsow U, Durham S, Fokkens W, Gjomarkaj M, Haahtela T, Bom AT, Wohrl S, Maibach H, Lockey R. The skin prick test - European standards. Clin Transl Allergy. 2013 Feb 1;3(1):3. doi: 10.1186/2045-7022-3-3. PMID 23369181
- [Background] Chaves C, de Andrade CR, Ibiapina C. Objective measures for functional diagnostic of the upper airways: practical aspects. Rhinology. 2014 Jun;52(2):99-103. doi: 10.4193/Rhino13.109. PMID 24932618
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Result] Orlandi RR, Smith TL, Marple BF, Harvey RJ, Hwang PH, Kern RC, Kingdom TT, Luong A, Rudmik L, Senior BA, Toskala E, Kennedy DW. Update on evidence-based reviews with recommendations in adult chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Jul;4 Suppl 1:S1-S15. doi: 10.1002/alr.21344. Epub 2014 May 29. PMID 24889751
- [Result] Baguley C, Brownlow A, Yeung K, Pratt E, Sacks R, Harvey R. The fate of chronic rhinosinusitis sufferers after maximal medical therapy. Int Forum Allergy Rhinol. 2014 Jul;4(7):525-32. doi: 10.1002/alr.21315. Epub 2014 Mar 7. PMID 24610673
- [Result] Watanabe S, Pinto JM, Bashir ME, De Tineo M, Suzaki H, Baroody FM, Naclerio RM, Sharma S. Effect of prednisone on nasal symptoms and peripheral blood T-cell function in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2014 Aug;4(8):609-16. doi: 10.1002/alr.21336. Epub 2014 Apr 21. PMID 24753507
- [Result] Poetker DM, Jakubowski LA, Lal D, Hwang PH, Wright ED, Smith TL. Oral corticosteroids in the management of adult chronic rhinosinusitis with and without nasal polyps: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Feb;3(2):104-20. doi: 10.1002/alr.21072. Epub 2012 Aug 7. PMID 22887970
- [Result] Lal D, Hwang PH. Oral corticosteroid therapy in chronic rhinosinusitis without polyposis: a systematic review. Int Forum Allergy Rhinol. 2011 Mar-Apr;1(2):136-43. doi: 10.1002/alr.20024. PMID 22287332